CLINICAL TRIAL: NCT00875667
Title: A Phase 2, Multicenter, Randomized Open-Label Study To Determine the Efficacy of Lenalidomide (Revlimid®) Versus Investigator's Choice in Patients With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: A Study to Determine the Efficacy of Lenalidomide Versus Investigator's Choice in Patients With Relapsed or Refractory Mantle Cell Lymphoma (MCL)
Acronym: Sprint
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MCL-002
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Mantle Cell Lymphoma; Lymphoma, Mantle-Cell
Keywords: Mantle Cell Lymphoma; Relapsed Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma; Lymphoma; MCL
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — Lenalidomide; Chlorambucil; Rituximab; Cytarabine; Gemcitabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide (Experimental): Lenalidomide
  Interventions: Drug: Lenalidomide
- Investigators choice single agent (Active Comparator): Investigators choice single agent - Chlorambucil, Rituximab, Cytarabine, Gemcitabine, Fludarabine
  Interventions: Drug: Investigators choice single agent

INTERVENTIONS:
Drug: Lenalidomide — For patients with a creatinine clearance of ≥ 60 mL/min: 25 mg daily x 21 days of a 28 day cycle until disease progression or unacceptable toxicity.
  For patients who have a moderate renal insufficiency (creatinine clearance is ≥ 30 mL/min but < 60mL/min: 10 mg daily x 21 days of a 28 day cycle (Cycles 1 and 2). After Cycle 2, if the patient remains free of Grade 3 or Grade 4 toxicity, the dose will be increased to 15 mg daily x 21 days of a 28 day cycle until disease progression or unacceptable toxicity.
  Other Names: Revlimid; Rev; CC-5013
  Arms: Lenalidomide
Drug: Investigators choice single agent — Investigators choice single agent - Chlorambucil, Rituximab, Cytarabine, Gemcitabine, or Fludarabine
  Other Names: Leukeran; Ritux; Rituxan; cytosine arabinoside; Ara-C; Cytosar-U; Gemzar; fludarabine phosphate; Fludara
  Arms: Investigators choice single agent

SUMMARY:
To evaluate the safety and efficacy of lenalidomide versus investigator choice in patients with relapsed or refractory mantle cell lymphoma.

DETAILED DESCRIPTION:
This research study is for patients who have relapsed or refractory mantle cell lymphoma following treatment such as radiotherapy, immunotherapy, chemotherapy, or radioimmunotherapy. Chemotherapy agents such as gemcitabine, cytarabine, chlorambucil, fludarabine, or the immunotherapeutic agent, rituximab, may be proposed. Thus, the aim is to search for new treatments that may improve the prognosis of patients with relapsed mantle cell lymphoma.

The present clinical study aims at determining if lenalidomide is safe and active in patients with mantle cell lymphoma who are refractory to their treatment or have relapsed once, twice or three times. Enrollment goal was met on March 7th 2013 and thus enrollment was stopped.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven mantle cell lymphoma
* Patients who are refractory to their regimen or have relapsed once, twice or up to three times and who have documented progressive disease
* Eastern Cooperative Oncology Group (ECOG) performance score 0,1, or 2
* Willing to follow pregnancy precaution

Exclusion Criteria:

* Any of the following laboratory abnormalities
* Absolute neutrophil count (ANC) < 1,500 cells/mm^3 (1.5 x 10^9/L)
* Platelet count < 60,000/mm^3 (60 x 10^9/L)
* Serum aspartate transaminase/serum glutamic oxaloacetic transaminase(AST/SGOT) or alanine transaminase/serum glutamic pyruvic transaminase (ALT/SGPT) >3.0 x upper limit or normal (ULN), except patients with documented liver involvement by lymphoma
* Serum total bilirubin > 1.5 x ULN, except in case of Gilbert's Syndrome and documented liver involvement by lymphoma.
* Calculated creatinine clearance (Cockcroft-Gault formula) of < 30 mL/min
* History of active central nervous system (CNS) lymphoma within the previous 3 months
* Subjects not willing to take deep venous thrombosis (DVT) prophylaxis
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are sero-positive because of hepatitis B virus vaccine are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2009-04-30 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marek Trneny, MD/PhD/Prof, Principal Investigator — Head, Ist Dept Medicine, Charles University Hospital; Director, Institute of Hematology and Blood Transfusion; Chair, Czech Lymphoma Study Group
Locations (97):
- Belgium (4):
  - UZ Brussels, Brussels
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - Cliniques Universitaires UCL de Mont-Godine, Yvoir
- Czechia (3):
  - Teaching Hospital BrnoHemato-oncology Dept, Brno
  - University Hospital2.Dep. of Int.med. hematology, Hradec Králové
  - Charles University General Hospital, Prague
- Denmark (2):
  - Rigshospitalet Department of Haematology L4042, Copenhagen
  - Herlev Hospital, Herlev
- France (20):
  - Polyclinique Bordeaux Nord Aquitaine Service Onco-Hematologie, Bordeaux
  - Hotel Dieu, Clermont-Ferrand
  - CHU Hopital Michallon, Grenoble
  - Centre Hospitalier Departemental Les Oudrairies, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - CHRU-Hopital Claude Huriez, Lille
  - CHU Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CHU Montpellier - Hôpital Saint Eloi, Montpellier
  - CHRU - Hotel Dieu, Nantes
  - Centre Antoine Lacassagne Oncologie medicale et Hematologie, Nice
  - Hopital Saint-Louis, Paris
  - CHRU - Hopital du Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Rennes Hematology, Rennes
  - Centre Henri Becquerel, Rouen
  - Hopital civil, Strasbourg
  - CHRU Hôpital de Hautepierre, Strasbourg
  - CHRU Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (9):
  - Uniklinik Koln, Cologne
  - Universitatsklinikum Essen, Essen
  - Universitaetsklinikum FreiburgInnere Med.1, Haematologie, Freiburg im Breisgau
  - UKG Universitatsklinikum Gottingen, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - Universitatsklinikum des Saarlandes, Homburg-Saar
  - Stadtisches Klinikum Karlsruhe, Karlsruhe
  - Universitatsklinik Munster, Münster
  - University of Ulm, Ulm
- Greece (2):
  - Attikon General University Hospital of Athens, Athens
  - University of Patras, Pátrai
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah University Hospital, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Italy (15):
  - A.O. Policlinico - Università di Bari, Bari
  - A.O.U. di Bologna Policlinico S.Orsola-Malpighi, Bologna
  - Ospedale Regionale di Bolzano, Bolzano
  - Ospedale Ferrarotto, Catania
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Ematologia ed Immunologia, Lecce
  - Istituto Europeo di Oncologia - IEO, Milan
  - San Raffaele Scientific Institute, Milan
  - Az. Osp. Vincenzo Cervello, Palermo
  - I.R.C.C.S. Policlinico San Matteo, Pavia
  - Az. Osp di Perugia, Perugia
  - Ospedale S. Chiara, Pisa
  - Azienda Ospedaliera "Bianchi-Melacrino-Morelli", Reggio Calabria
  - Reference Cancer Center of Basilicata, Rionero in Vulture
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Netherlands (3):
  - Meander Medisch Centrum, Amersfoort
  - Medisch Spectrum Twente, Enshede
  - Isala Klinieken, Zwolle
- Poland (6):
  - Malopolskie Centrum medyczne s.c., Krakow
  - Uniwersytet Jagiellonski Collegium Medicum, Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi, Lodz
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie w Warszawie, Warsaw
  - Nowotworww Krwi i Transplantacji Szpiku, Wroclaw
  - Dolnoslaskie Centrum Transplantacji Komorkowych, Wroclaw
- Russia (13):
  - Republic Clinical Oncology Dispensary, Kazan'
  - Institution of Russian Academy of Medical Sciences Russian Oncological Research Centre n.a. N. N. Bl, Moscow
  - Nizhegorodskiy Regional Clinical Hospital named after N.A. Semashko, Nizhny Novgorod
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Medical Radiology Research Centre RAMS, Obninsk
  - Perm Territorial Oncology Dispensary, Perm
  - Scientific Research Institute of OncologySoft Tissue Department, Rostov-on-Don
  - St. Petersburg Research Institute of Hematology and Blood Transfusion, Saint Petersburg
  - St. Petersburg Pavlov State Medical University, Saint Petersburg
  - Federal Centre of Heart, Blood and Endocrinology of Rosmed technlologies V.A. Almazov, Saint Petersburg
  - Saratov Medical University Chair of Professional Pathology and Haematology, Saratov
  - Volgograd Regional Clinical Oncology Dispensary 1, Volgograd
  - Sverdlovsk Regional Clinical Hospital 1, Yekaterinburg
- Spain (5):
  - Hospital Universitario Vall D Hebron, Barcelona
  - Hospital de La Princesa, Madrid
  - Hospital La Paz, Madrid
  - Hospital Costa del Sol, Marbella
  - Clinica Universitaria de Navarra, Pamplona
- Sweden (2):
  - Lund University Hosptial, Lund
  - University Hospital Uppsala, Uppsala
- United Kingdom (9):
  - Royal Bournemouth Hosp, Bournemouth
  - Addenbrookes Hospital, Cambridge
  - Royal Liverpool University Hospital, Liverpool
  - Christie Hospital, Manchester
  - Newcastle Hospital Foundation Trust, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton
  - The Royal Wolverhampton Hospital NHS Trust, Wolverhampton

REFERENCES:
- [Background] Trneny M, Lamy T, Walewski J, Belada D, Mayer J, Radford J, Jurczak W, Morschhauser F, Alexeeva J, Rule S, Afanasyev B, Kaplanov K, Thyss A, Kuzmin A, Voloshin S, Kuliczkowski K, Giza A, Milpied N, Stelitano C, Marks R, Trumper L, Biyukov T, Patturajan M, Bravo MC, Arcaini L; SPRINT trial investigators and in collaboration with the European Mantle Cell Lymphoma Network. Lenalidomide versus investigator's choice in relapsed or refractory mantle cell lymphoma (MCL-002; SPRINT): a phase 2, randomised, multicentre trial. Lancet Oncol. 2016 Mar;17(3):319-331. doi: 10.1016/S1470-2045(15)00559-8. Epub 2016 Feb 16. PMID 26899778
- [Derived] Hagner PR, Chiu H, Ortiz M, Apollonio B, Wang M, Couto S, Waldman MF, Flynt E, Ramsay AG, Trotter M, Gandhi AK, Chopra R, Thakurta A. Activity of lenalidomide in mantle cell lymphoma can be explained by NK cell-mediated cytotoxicity. Br J Haematol. 2017 Nov;179(3):399-409. doi: 10.1111/bjh.14866. Epub 2017 Aug 2. PMID 28771673

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 67 sites including 3 sites in Belgium, 3 in Czech Republic, 14 in France, 7 in Germany, 2 in Israel, 10 in Italy, 1 in the Netherlands, 5 in Poland, 11 in Russia, 4 in Spain, 2 in Sweden, and 5 in the United Kingdom (UK).
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive lenalidomide monotherapy or investigator's choice. Participants were stratified according to the time since diagnosis (< 3 years or ≥ 3 years), time since last treatment (< 6 months [refractory] or ≥ 6 months) and if they had undergone a prior stem cell transplant or not.
Groups:
- Lenalidomide: Participants received lenalidomide 25 mg capsules orally every day for 21 days of each 28-day treatment cycle until disease progression or unacceptable toxicity. Participants with moderate renal insufficiency (creatinine clearance is ≥ 30 mL/min but < 60mL/min received 10 mg lenalidomide for 21 days of each 28-day cycle (Cycles 1 and 2). After Cycle 2, if the participant remained free of Grade 3 or Grade 4 toxicity, the dose was increased to 15 mg lenalidomide for 21 days of each 28-day treatment cycle until disease progression or unacceptable toxicity.
- Investigators Choice: Participants received a single agent investigators choice (IC) of chlorambucil 40 mg/m^2 PO every 28 days until progressive disease (PD) or toxicity, OR rituximab 375 mg/m^2 by intravenous (IV) infusion on days 1, 8, 15 and 22 of each 56-day treatment cycle until PD or toxicity, OR cytarabine 1-2 g/m^2 by IV infusion on days 1 and 2 of each 28 day treatment cycle; up to 6 cycles, OR gemcitabine 1000 mg/m^2 by IV infusion on days 1, 8 and 15 of each 28 day treatment cycle; up to 6 cycles OR oral fludarabine 40 mg/m^2 or IV fludarabine 25 mg/m^2 on days 1 through 5 of each 28-day cycle; up to 6 cycles. Participants were given the option to enter into the lenalidomide crossover phase if PD occurred and received lenalidomide 25 mg capsules daily on days 1 to 21 of each 28 day treatment cycle until PD or toxicity.
Period: Overall Study
Arm/Group | Lenalidomide | Investigators Choice
Started | 170 | 84
Crossover From IC to Lenalidomide (Upon disease progression, participants crossed over to lenalidomide) | 0 (NA = Participants in the IC arm were able to crossover to lenalidomide) | 40 (Upon disease progression, participants crossed over to lenalidomide)
Participants Treated | 167 | 83
Completed | 0 | 11 (Participants completed 6 cycles of IC single agent cytarabine, fludarabine, or gemcitabine.)
Not Completed | 170 | 73
Not completed — Adverse Event | 29 | 10
Not completed — Withdrawal by Subject | 17 | 5
Not completed — Death | 7 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Disease Progression | 100 | 49
Not completed — Miscellaneous | 12 | 6
Not completed — Randomized but no Study Drug Given | 3 | 1

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population was defined as all participants who were randomized, independent of whether they received study treatment or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide | Investigators Choice | Total
Number analyzed (Participants) | 170 | 84 | 254
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (9.38) | 67.5 (8.20) | 67.8 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 21 | 68
  Male | 123 | 63 | 186
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 161 | 80 | 241
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 4 | 13
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a subject's disease is progressing, assess how the disease affects the daily living activities of the subject and determine appropriate treatment and prognosis. 0 = Fully Active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out light work; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities; 3 = Capable of only limited self-care; 4 = Completely Disabled, No self-care
  Participants
    0 = Fully Active | 65 | 36 | 101
    1 = Restrictive but Ambulatory | 77 | 37 | 114
    2 = Ambulatory but Unable to Work | 27 | 11 | 38
    3 = Limited Self-Care | 0 | 0 | 0
    Missing | 1 | 0 | 1
Stage of Mantle Cell Lymphoma (MCL) at Diagnosis [Count of Participants; unit: Participants] — Ann Arbor staging is the staging system for lymphomas, both in Hodgkin's lymphoma (previously called Hodgkin's disease) and Non-Hodgkin lymphoma (abbreviated NHL). Stage I = Involvement of 1 Lymph Node (LN) or extralymphatic region Stage II = ≥ 2 LN sites on the same side of the diaphragm Stage III = LN regions on both sides of the diaphragm; may include spleen and 1 extralymphatic organ Stage IV = involvement of ≥ 1 extralymphatic organs with or without associated LN involvement (diffuse or disseminated)
  Participants
    Stage I | 3 | 2 | 5
    Stage II | 10 | 1 | 11
    Stage III | 30 | 20 | 50
    Stage IV | 123 | 59 | 182
    Missing | 4 | 2 | 6
MCL International Prognostic Index (MIPI) Score at Baseline [Count of Participants; unit: Participants] — A prognostic index predictive of the outcome in advanced mantle cell lymphoma
  Participants
    Low Risk | 42 | 21 | 63
    Intermediate Risk | 66 | 37 | 103
    High Risk | 60 | 25 | 85
    Missing | 2 | 1 | 3
Bone Marrow Involvment as Baseline [Count of Participants; unit: Participants] — Bone marrow involvement (biopsy score) was categorized according to the following observations (Cheson, 1999):
  (i) positive, if unequivocal cytologic or architectural evidence of malignancy, (ii) negative, if no aggregates or only a few well-circumscribed lymphoid aggregates, or (iii) indeterminate, if increased number or size of aggregates without cytologic or architectural atypia
  Participants
    Negative | 27 | 11 | 38
    Intermediate | 4 | 3 | 7
    Positive | 21 | 13 | 34
    Missing | 118 | 57 | 175

OUTCOME MEASURES:

1. Primary Outcome: Kaplan Meier Estimate for Progression Free Survival (PFS) by Independent Review Committee (IRC) Central Review
Description: PFS was defined as time of randomization to the first observation of disease progression or death due to any cause, whichever was first. If a participant had not progressed or died, PFS was censored at the time of last assessment when the participant was known not to have progressed. For participants who received other anti-lymphoma therapy with no evidence of progression, PFS was censored at time of last tumor assessment with no evidence of progression prior to the start of new anti-lymphoma treatment.
Time Frame: From randomization to progression of disease or death; up to data cut off date of 07 March 2014; overall median follow-up time was 93.9 weeks
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
weeks | 37.6 [24.0 to 52.6] | 22.7 [15.9 to 30.1]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.012, Stratified Log Rank Test — Stratification factors were: time from diagnosis to first dose, time from last prior anti-lymphoma therapy to first dose, prior stem cell transplant, and MIPI at baseline; Stratified Hazard Ratio = 0.63, 95% CI 2-sided [0.43 to 0.90]

2. Primary Outcome: Kaplan Meier Estimate for Progression Free Survival by Investigator's Assessment at the Final Analysis
Description: Kaplan Meier estimates of PFS were defined as the time from randomization to the first observation of disease progression or death due to any cause, whichever was first. If a participant had not progressed or died, PFS was censored at the time of last completed assessment when the participant was known not to have progressed. For participants who received other anti-lymphoma therapy with no evidence of progression, PFS was censored at time of last tumor assessment with no evidence of progression prior to the start of new anti-lymphoma treatment.
Time Frame: From randomization to progression of disease or death; up to study discontinuation of 09 October 2018; overall median follow-up time was 285 weeks
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
weeks | 37.3 [24.1 to 52.6] | 23.6 [15.9 to 33.3]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.003, Stratified Log Rank Test — [p-value comment as in outcome 1, analysis 1]; Stratified Hazard Ratio = 0.60, 95% CI 2-sided [0.43 to 0.85] — The weights are based on observed events at the time the third DMC meeting was held and based on the difference between observed and expected events at the time of the primary analysis

3. Secondary Outcome: Percentage of Participants Who Achieved an Overall Response According to the IRC Central Review
Description: Overall Response Rate (ORR) was defined as the percentage of participants whose best response was Complete Response (CR), Complete Response unconfirmed (CRu) or Partial Response (PR). Participants who discontinued before any response had been observed or changed to other anti-lymphoma treatments before response had been observed, were considered as non-responders. Tumor Response was assessed by a modification of the International Lymphoma Workshop Response Criteria, IWRC, Cheson, 1999; CR is defined as the disappearance of all clinical and radiographic evidence of disease; CRu is defined as a CR, with a 1) residual lymph node mass >1.5 cm that has decreased by 75% in the sum of the product of the diameters (SPD). Individual nodes previously confluent decreased by more than 75% in the SPD compared with original mass; 2) indeterminate bone marrow; PR = is defined ≥50% decrease in 6 largest nodes or nodal masses.
Time Frame: From date of randomization to the data cut-off date of 07 March 2014; median treatment duration was 24.3 weeks for the lenalidomide arm and 13.1 weeks for the investigators choice arm
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
Percentage of Participants | 40.0 [32.58 to 47.78] | 10.7 [5.02 to 19.37]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p < 0.001, Chi-squared

4. Secondary Outcome: Percentage of Participants Who Achieved an Overall Response as Assessed by the Investigator at the Final Analysis
Description: Overall Response Rate (ORR) was defined as the percentage of participants whose best response was Complete Response, Complete Response unconfirmed or Partial Response. Participants who had discontinued before any response has been observed or changed to other anti-lymphoma treatments before response had been observed, were considered as non-responders. Tumor Response was assessed by a modification of the International Lymphoma Workshop Response Criteria, IWRC, Cheson, 1999; CR is defined as the disappearance of all clinical and radiographic evidence of disease; CRu is defined as a CR, with a 1) residual lymph node mass >1.5 cm that has decreased by 75% in the sum of the product of the diameters (SPD). Individual nodes previously confluent decreased by more than 75% in the SPD compared with original mass; 2) indeterminate bone marrow; PR = is defined ≥50% decrease in 6 largest nodes or nodal masses.
Time Frame: From date of randomization to the study discontinuation date of 09 October 2018; median treatment duration was 24.3 weeks for lenalidomide and 13.1 weeks for the investigator choice arm
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
Percentage of Participants | 45.9 [38.23 to 53.68] | 22.6 [14.20 to 33.05]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p < 0.001, Chi-squared

5. Secondary Outcome: Kaplan Meier Estimate for Duration of Response (DOR) According to the IRC Central Review
Description: Duration of response was defined as the time from when the first response of CR, CRu, or PR was first achieved until documented tumor progression, or until the participant died from any cause, whichever occurred first. Participants who did not progress or die at the time of analysis were censored at the last assessment date that the participant was known to be progression-free. Participants who received a new treatment without documented progression were censored at the last assessment date that the participant was known to be progression-free.
Time Frame: From date of randomization to the data cut-off date of 07 March 2014; median study duration was 70.7 weeks for the lenalidomide arm and 69.3 weeks for the investigators choice arm
Population: The analysis population included participants with an overall response.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 68 | 9
Weeks | 69.6 [41.1 to 86.7] | 45.1 [36.3 to 80.9]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.421, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.29 to 1.68]

6. Secondary Outcome: Kaplan Meier Estimate for Duration of Response as Assessed by the Investigator at the Final Analysis
Description: as for outcome 5
Time Frame: From date of randomization to the study discontinuation date of 09 October 2018; median study duration was 103.9 weeks for lenalidomide and 87.0 weeks for the investigator choice arm
Population: The analysis population included participants with an overall response.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 78 | 19
Weeks | 70.1 [47.0 to 98.0] | 91.7 [28.3 to 130.1]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.875, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.52 to 1.74]

7. Secondary Outcome: Percentage of Participants With a Complete Response, Unconfirmed Complete Response, Partial Response and Stable Disease According to the IRC Central Review
Description: Tumor control rate was defined as the percentage of participants with a complete response (CR), unconfirmed complete response (CRu), partial response (PR) and stable disease (SD). Tumor Response was assessed by a modification of the International Lymphoma Workshop Response Criteria, IWRC, Cheson, 1999); CR is defined as the disappearance of all clinical and radiographic evidence of disease; CRu is defined as a CR, with a 1) residual lymph node mass >1.5 cm that has decreased by 75% in the sum of the product of the diameters (SPD). Individual nodes previously confluent decreased by more than 75% in the SPD compared with original mass; 2) indeterminate bone marrow; PR = is defined ≥50% decrease in 6 largest nodes or nodal masses. Stable disease (SD) is defined as less than a PR (see above) but is not progressive disease or relapsed disease.
Time Frame: as for outcome 3
Population: ITT population includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
Percentage of Participants | 69.4 [61.89 to 76.24] | 63.1 [51.87 to 73.37]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.313, Chi-squared

8. Secondary Outcome: Percentage of Participants With a Complete Response, Unconfirmed Complete Response, Partial Response and Stable Disease at the Final Analysis
Description: as for outcome 7
Time Frame: From date of randomization to the discontinuation date of 09 October 2018; median treatment duration was 24.3 weeks for the lenalidomide arm and 13.1 weeks for the investigators choice arm
Population: ITT population includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
Percentage of participants | 70.0 [62.51 to 76.78] | 65.5 [54.31 to 75.52]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.465, Chi-squared

9. Secondary Outcome: Kaplan Meier Estimate of Time to Progression According to the IRC Central Review
Description: Time to progression (TTP) was defined as the time from randomization until objective tumor progression. Time to progression did not include deaths. Participants without progression at the time of analysis were censored at the last assessment date that the participant was known to be progression-free. Participants who received a new anti-lymphoma treatment without documented progression were censored at the last assessment date that the participant was known to be progression-free.
Time Frame: as for outcome 5
Population: ITT population includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
Weeks | 39.3 [24.3 to 52.9] | 24.7 [15.9 to 30.1]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.005, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.45 to 0.87]

10. Secondary Outcome: Kaplan Meier Estimate of Time to Progression as Assessed by the Investigator at the Final Analysis
Description: as for outcome 9
Time Frame: as for outcome 6
Population: ITT population includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
Weeks | 39.3 [25.1 to 61.0] | 24.7 [15.9 to 36.7]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.003, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.46 to 0.86]

11. Secondary Outcome: Kaplan Meier Estimate of Time to Treatment Failure (TTF) as Assessed by the Investigator
Description: Time to treatment failure was defined as the time from the first dose of study drug to discontinuation of treatment for any reason, including disease progression assessed by the investigator, treatment toxicity, or death. Participants who were on-treatment or completed the treatment according to the protocol were censored at the last date of drug intake.
Time Frame: From the date of the first treatment to the data cut-off date of 07 March 2014; median treatment duration was 24.3 weeks for the lenalidomide arm and 13.1 weeks for the investigators choice arm
Population: Includes all treated participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 167 | 83
weeks | 24.4 [17.1 to 37.6] | 17.9 [14.1 to 24.9]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.046, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.54 to 1.00]

12. Secondary Outcome: Kaplan Meier Estimate of Time to Treatment Failure as Assessed by the Investigator at the Final Analysis
Description: as for outcome 11
Time Frame: From date of first dose of treatment to the study discontinuation date of 09 October 2018; median treatment duration was 24.3 weeks for lenalidomide and 13.1 weeks for the investigator choice arm
Population: Includes all treated participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 167 | 83
weeks | 24.4 [17.1 to 37.6] | 17.9 [14.1 to 24.9]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.095, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.58 to 1.05]

13. Secondary Outcome: Kaplan Meier Estimate of Time to First Response (TTFR) According to the IRC Central Review
Description: Time to Response was defined as the time from first dose of study drug to the date of the first response (having at least a PR) and was calculated only for responding participants. ). Participants with progression at the time of analysis were censored at the first assessment date that the participant was known to have progressed. Participants with SD at the time of analysis were censored at the last assessment date that the participant was known to be progression-free.
Time Frame: From randomization of study drug to time of first documented PR or better response; up to data cut-off date of 07 March 2014; median treatment duration was 24.3 weeks for the lenalidomide arm and 13.1 weeks for the investigators choice arm
Population: ITT population includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
Weeks | 18.7 [16.7 to 49.7] | NA [63.9 to NA] — Not estimable due to the low number of participants with a response.
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 3.91, 95% CI 2-sided [1.95 to 7.85]

14. Secondary Outcome: Kaplan Meier Estimate of Time to First Response as Assessed by the Investigator at the Final Analysis
Description: Time to first response was defined as the time from first dose of study drug to the date of the first response (having at least a PR). Participants with progression at the time of analysis were censored at the first assessment date that the participant was known to have progressed. Participants with SD at the time of analysis were censored at the last assessment date that the subject was known to be progression-free.
Time Frame: as for outcome 4
Population: ITT population includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
Weeks | 23.9 [16.7 to 25.6] | 40.0 [25.6 to NA] — Upper Limit not estimable due to the low number of participants with a response.
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p < 0.004, Log Rank; Hazard Ratio (HR) = 2.06, 95% CI 2-sided [1.24 to 3.42]

15. Secondary Outcome: Kaplan Meier Estimate for Overall Survival (OS) According to the IRC Central Review
Description: Overall survival was defined as the time from randomization until death from any cause. Participants alive or lost to follow-up at the time of analysis were censored at the last date they were known to be alive.
Time Frame: From date of randomization to the data cut-off date of 07 March 2014; overall median follow-up was 93.9 weeks
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
weeks | 121.0 [86.7 to 160.4] | 91.7 [69.4 to 125.6]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.519, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.62 to 1.28]

16. Secondary Outcome: Kaplan Meier Estimate for Overall Survival as Assessed by the Investigator at the Final Analysis
Description: as for outcome 15
Time Frame: From randomization to progression of disease or death; up to the study discontinuation date of 09 October 2018; overall median follow-up time was 285 weeks
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 170 | 84
weeks | 120.6 [98.1 to 153.0] | 91.7 [69.4 to 137.3]
Statistical Analysis 1: Comparison: Lenalidomide vs Investigators Choice; Test type: Superiority; p = 0.558, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.67 to 1.25]

17. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Adverse events were assessed using National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 3: according to the following scale: Grade 1 = Mild Adverse Event (AE), Grade 2 = Moderate AE, Grade 3 = Severe and Undesirable AE, Grade 4 = Life-threatening or Disabling AE, and Grade 5 = Death; Serious AEs (SAEs) are those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes listed above. after the first dose of study drug and within 28 days after the last dose. A Treatment Emergent Adverse event (TEAE) is defined as any AE occurring or worsening on or after the first dose of study drug and within 28 days after the last dose of study drug.
Time Frame: From the date of the first dose of study drug to 28 days after the last dose, up to the study discontinuation date of 09 October 2018; median treatment duration was 24.3 weeks for lenalidomide and 13.1 weeks for the investigators choice arm
Population: The safety population included participants who received at least one dose of study drug (either lenalidomide or investigator's choice).
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 167 | 83
Participants
  Any TEAE | 159 | 69
  Any TEAE Grade 3 AE | 126 | 49
  Any TEAE Grade 4 AE | 56 | 29
  Any TEAE Grade 5 AE | 15 | 2
  Any TEAE Related to the IP | 141 | 51
  Any Grade 3 AE Related to IP | 106 | 36
  Any Grade 4 AE Related to IP | 46 | 19
  Any Grade 5 AE Related to IP | 0 | 0
  Any Serious Adverse Event (SAE) | 75 | 22
  Any SAE Related to IP | 38 | 12
  Any TEAE Leading to Stopping of IP | 31 | 14
  Any Treatment Related AE Leading to Stopping IP | 18 | 7
  TEAE Leading to Dose Reduction/Interruption | 114 | 33
  Related AE Leading to Dose Reduct/Interruption | 103 | 29
  TEAE Leading to Dose Reduction | 72 | 13
  Related AE Leading to Dose Reduction | 69 | 10
  TEAE Leading to Dose Interruption | 110 | 28
  Related AE Leading to Dose Interruption | 98 | 25

18. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Physical Functioning Domain
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Physical Functioning Scale ranges from 0 to 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Baseline known as screening visit, after cycle 2 (C3D1), after Cycle 4 (C5D1), after Cycle 6, (C7D1), after Cycle 8, (C9D1) and at discontinuation; median treatment duration was 24.3 weeks for lenalidomide and 13.1 weeks for the investigator choice arm.
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale
  Baseline | 71.8 (22.35) | 78.9 (17.38)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 104 | 43
  Change from Baseline to Cycle 3 Day 1 | -0.5 (15.47) | -3.7 (16.22)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 70 | 26
  Change from Baseline to Cycle 5 Day 1 | 1.6 (15.18) | -2.1 (19.02)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 56 | 8
  Change from Baseline to Cycle 7 Day 1 | 2.4 (16.74) | 4.2 (16.69)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 46 | 6
  Change from Baseline to Cycle 9 Day 1 | 2.8 (18.08) | 11.1 (11.67)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | -5.6 (19.46) | -5.1 (17.14)

19. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Physical Functioning Domain to Treatment Discontinuation Visit
Description: as for outcome 18
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 124 | 57
units on a scale | 3.4 (18.70) | -1.8 (17.57)

20. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Role Functioning Domain
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Role Functioning Scale ranges from 0 to 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale
  Baseline | 71.5 (31.10) | 73.9 (25.60)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | -4.8 (26.12) | 3.5 (21.69)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | 1.4 (26.09) | -6.4 (30.21)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Change from Baseline to Cycle 7 Day 1 | 0.3 (26.44) | 0.0 (38.83)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | 1.8 (26.75) | 13.9 (19.48)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | -9.1 (29.05) | -4.3 (31.09)

21. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Role Functioning Domain to Treatment Discontinuation Visit
Description: as for outcome 20
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale | 3.1 (28.43) | 5.0 (27.09)

22. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Cognitive Functioning Domain
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Cognitive Functioning Domain ranges from 0 to 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale
  Baseline | 84.6 (19.86) | 83.6 (20.18)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | 0.0 (16.34) | -2.3 (13.89)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | -1.9 (17.72) | 1.3 (14.85)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Change from Baseline to Cycle 7 Day 1 | -3.2 (19.27) | 4.2 (14.77)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | -2.5 (18.05) | 5.6 (13.61)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | -5.1 (19.46) | -2.3 (15.68)

23. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Cognitive Functioning Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Cognitive Functioning Scale ranges from 0 to 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale | 3.2 (17.92) | 2.9 (14.13)

24. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Social Functioning Domain
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Social Functioning Domain ranges from 0 to 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale
  Baseline | 74.9 (28.39) | 78.4 (26.85)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | -1.0 (20.39) | -1.2 (22.54)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | 1.6 (19.75) | -4.5 (29.27)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Change from Baseline to Cycle 7 Day 1 | -1.5 (25.06) | 2.1 (28.78)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | 4.3 (22.11) | 0.0 (23.57)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | -5.1 (24.63) | -2.7 (20.87)

25. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Social Functioning Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Social Functioning Scale ranges from 0 to 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale | 5.1 (20.87) | 3.8 (19.92)

26. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Fatigue Domain
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Fatigue Domain was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale
  Baseline | 40.2 (26.67) | 39.2 (23.50)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | 0.1 (21.72) | 2.1 (22.12)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | -3.2 (20.84) | 3.4 (25.68)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Change from Baseline to Cycle 7 Day 1 | -1.0 (21.03) | -6.9 (25.85)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | -3.9 (26.64) | -7.4 (25.01)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | 5.2 (21.48) | 2.6 (24.11)

27. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Fatigue Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Fatigue Scale was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale | -4.9 (22.76) | -2.9 (23.24)

28. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Pain Domain
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Pain Domain was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale
  Baseline | 22.6 (25.86) | 13.7 (20.15)
  Cycle 3 Day 1: number analyzed (Participants) | 104 | 43
  Cycle 3 Day 1 | -2.2 (19.99) | -1.2 (25.30)
  Cycle 5 Day 1: number analyzed (Participants) | 70 | 26
  Cycle 5 Day 1 | -0.2 (24.82) | -2.6 (20.38)
  Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Cycle 7 Day 1 | 3.2 (26.99) | 0.0 (19.92)
  Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Cycle 9 Day 1 | -3.2 (25.92) | -2.8 (6.80)
  Treatment Discontinuation: number analyzed (Participants) | 61 | 43
  Treatment Discontinuation | 4.6 (26.38) | 3.5 (22.29)

29. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Pain Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Pain Scale was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: Baseline known as screening visit, after cycle 2 (C3D1), after Cycle 4 (C5D1), after Cycle 6, (C7D1), after Cycle 8, (C9D1) and time of discontinuation from treatment visit.Up to final data cut-0ff date of 07 March 2014
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale | -5.8 (24.61) | -3.5 (21.30)

30. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Nausea / Vomiting Domain
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Nausea and Vomiting Domain was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale
  Baseline | 4.9 (10.31) | 3.8 (11.22)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | 2.5 (14.39) | 0.4 (10.60)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | 2.6 (11.83) | 5.8 (21.57)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Change from Baseline to Cycle 7 Day 1 | 5.3 (17.30) | 2.1 (22.60)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | -0.7 (10.40) | 2.8 (6.80)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | 0.5 (9.99) | 6.6 (18.59)

31. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Nausea and Vomiting Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Nausea and Vomiting Scale was scored between 0 and 100, with a high score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale | -2.3 (8.82) | -0.6 (8.31)

32. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Constipation
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Constipation Domain was scored between 0 and 100, with a high score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale
  Baseline | 12.5 (23.27) | 8.6 (19.16)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | 6.3 (27.38) | -0.8 (18.53)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | 4.2 (25.78) | 1.3 (17.59)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Change from Baseline to Cycle 7 Day 1 | 3.5 (27.95) | 0.0 (30.86)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | -0.7 (20.25) | 0.0 (21.08)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | 10.2 (32.27) | 0.8 (21.19)

33. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Constipation Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Constipation Scale was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale | -0.3 (27.60) | -3.5 (16.29)

34. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Diarhoea
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Diarhoea Domain was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale
  Baseline | 15.7 (27.15) | 12.6 (20.42)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | -3.5 (25.71) | -3.1 (21.60)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | -4.2 (29.78) | 1.3 (22.07)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 55 | 8
  Change from Baseline to Cycle 7 Day 1 | 2.4 (32.62) | -4.2 (33.03)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | -2.1 (22.42) | 0.0 (36.51)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | 1.6 (30.44) | 0.0 (25.20)

35. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Diarhoea Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact).
  The EORTC QLQ-C30 Diarhoea Scale was scored between 0 and 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: as for outcome 29
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale | -7.2 (25.25) | -5.8 (21.93)

36. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Insomnia Domain
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Insomnia Domain was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale
  Baseline | 29.4 (30.69) | 25.7 (27.34)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | -7.6 (27.06) | -4.7 (31.36)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | -5.2 (24.97) | -6.4 (32.69)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Change from Baseline to Cycle 7 Day 1 | -1.8 (29.83) | -16.7 (39.84)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | -7.1 (30.25) | -16.7 (40.82)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | -3.2 (28.76) | 0.8 (22.41)

37. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Insomnia Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Insomnia Scale was scored between 0 and 100, with a high score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale | -12.8 (28.64) | -7.6 (30.87)

38. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Dyspnoea Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Dyspnoea Domain was scored between 0 and 100, with a high score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale
  Baseline | 26.5 (28.98) | 21.2 (28.97)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 103 | 43
  Change from Baseline to Cycle 3 Day 1 | -1.6 (27.76) | -0.8 (29.54)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 70 | 26
  Change from Baseline to Cycle 5 Day 1 | -1.4 (26.88) | 0.0 (33.99)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Change from Baseline to Cycle 7 Day 1 | -2.9 (25.42) | 4.2 (48.59)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | 1.4 (31.05) | 5.6 (25.09)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 61 | 43
  Change from Baseline to Treatment Discontinuation | 6.0 (28.22) | 0.8 (23.56)

39. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Dyspnoea Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Dyspnoea Domain to Treatment Scale was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale | -7.3 (25.70) | -5.8 (27.55)

40. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Appetite Loss Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Appetite Loss Domain was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale
  Baseline | 18.1 (27.69) | 16.2 (26.02)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | 2.5 (31.25) | -0.8 (34.49)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | 1.9 (28.67) | 5.1 (43.91)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Change from Baseline to Cycle 7 Day 1 | -2.3 (23.45) | -12.5 (46.93)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | -4.3 (27.47) | -11.1 (27.22)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | 4.8 (32.42) | 5.4 (27.15)

41. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Appetite Loss Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Appetite Loss Domain to Treatment Scale was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale | -4.8 (28.30) | -4.1 (29.59)

42. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Financial Problems Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Financial Problems Domain was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale
  Baseline | 19.5 (27.78) | 10.8 (19.98)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | -7.0 (25.61) | -0.8 (18.53)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | -7.0 (27.55) | -3.8 (23.71)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Change from Baseline to Cycle 7 Day 1 | -2.9 (33.50) | -4.2 (11.79)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | -9.2 (31.62) | -5.6 (13.61)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | -4.3 (22.97) | 1.6 (19.18)

43. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Financial Problems Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Financial Problems Domain Scale was scored between 0 and 100, with a higher score representing worse symptomatic expression.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale | -10.9 (25.32) | -2.3 (19.78)

44. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Global Health Status / QoL Domain
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Global Health Status / QoL Domain was scored between 0 and 100, with a higher score representing a higher quality of life.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale
  Baseline | 59.0 (21.45) | 58.4 (18.58)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | -3.4 (21.89) | 2.3 (18.66)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | -0.7 (19.96) | 3.2 (24.50)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 57 | 8
  Change from Baseline to Cycle 7 Day 1 | 1.0 (17.04) | 7.3 (29.36)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | 4.3 (21.76) | 8.3 (22.97)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | -5.8 (18.76) | -1.0 (19.26)

45. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Global Health Status / QoL Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Global Health Status / QoL Domain to Treatment Scale was scored between 0 and 100, with a higher score representing a higher quality of life.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale | 4.6 (19.06) | 5.6 (20.43)

46. Secondary Outcome: Mean Change From Baseline in the EORTC QLQ-C30 Emotional Functioning Domain
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Emotional Domain ranges from 0 to 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 161 | 74
units on a scale
  Baseline | 73.7 (21.52) | 78.5 (18.56)
  Change from Baseline to Cycle 3 Day 1: number analyzed (Participants) | 105 | 43
  Change from Baseline to Cycle 3 Day 1 | 3.4 (19.64) | 1.3 (20.77)
  Change from Baseline to Cycle 5 Day 1: number analyzed (Participants) | 71 | 26
  Change from Baseline to Cycle 5 Day 1 | 3.6 (17.01) | 1.3 (16.11)
  Change from Baseline to Cycle 7 Day 1: number analyzed (Participants) | 56 | 8
  Change from Baseline to Cycle 7 Day 1 | 8.1 (20.53) | -3.1 (26.33)
  Change from Baseline to Cycle 9 Day 1: number analyzed (Participants) | 47 | 6
  Change from Baseline to Cycle 9 Day 1 | 4.5 (21.96) | 1.4 (13.35)
  Change from Baseline to Treatment Discontinuation: number analyzed (Participants) | 62 | 43
  Change from Baseline to Treatment Discontinuation | -1.3 (22.05) | -1.5 (16.50)

47. Secondary Outcome: Maximum Change From Baseline in the EORTC QLQ-C30 Emotional Functioning Domain to Treatment Discontinuation Visit
Description: The EORTC-QLQ-C30 is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Emotional Functioning Scale ranges from 0 to 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: as for outcome 18
Population: Health Related Quality of Life (QoL) Evaluable Population includes participants who had evaluable QoL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Investigators Choice
Number analyzed (Participants) | 160 | 74
units on a scale | 6.9 (21.79) | 3.7 (17.11)

ADVERSE EVENTS:
Time Frame: From randomization of study drug to 30 days post-last dose; up to the study discontinuation date of 09 October 2018; median treatment duration was 24.3 weeks for lenalidomide and 13.1 weeks for the investigators choice arm.
Groups:
- Investigator's Choice: Participants received a single agent investigators choice (IC) of chlorambucil 40 mg/m^2 PO every 28 days until progressive disease (PD) or toxicity, OR rituximab 375 mg/m^2 by intravenous (IV) infusion on days 1, 8, 15 and 22 of each 56-day treatment cycle until PD or toxicity, OR cytarabine 1-2 g/m^2 by IV infusion on days 1 and 2 of each 28 day treatment cycle; up to 6 cycles, OR gemcitabine 1000 mg/m^2 by IV infusion on days 1, 8 and 15 of each 28 day treatment cycle; up to 6 cycles OR oral fludarabine 40 mg/m^2 or IV fludarabine 25 mg/m^2 on days 1 through 5 of each 28-day cycle; up to 6 cycles. Participants were given the option to enter into the lenalidomide crossover phase if PD occurred and received lenalidomide 25 mg capsules daily on days 1 to 21 of each 28 day treatment cycle until PD or toxicity.
Arm/Group | Lenalidomide | Investigator's Choice
All-Cause Mortality (participants affected / at risk) | 119/167 | 59/83
Serious Adverse Events (participants affected / at risk) | 75/167 | 22/83
Other Adverse Events (participants affected / at risk) | 146/167 | 61/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=167) | Investigator's Choice (N=83)
ANAEMIA (Blood and lymphatic system disorders) | 6 | 2
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 6 | 2
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 1 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 6 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 2
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 2 | 0
CARDIAC FAILURE (Cardiac disorders) | 2 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0
DEAFNESS BILATERAL (Ear and labyrinth disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 6 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 2 | 0
DEATH (General disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3 | 1
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 2 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PYREXIA (General disorders) | 5 | 2
SUDDEN DEATH (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 0
ASPERGILLUS INFECTION (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 2 | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 1
LUNG INFECTION (Infections and infestations) | 2 | 0
MENINGITIS VIRAL (Infections and infestations) | 1 | 0
NEUTROPENIC SEPSIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 6 | 3
PNEUMONIA MORAXELLA (Infections and infestations) | 0 | 1
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1 | 0
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 0
SINUSITIS (Infections and infestations) | 1 | 0
SKIN INFECTION (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0
UROSEPSIS (Infections and infestations) | 1 | 0
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 1
WEIGHT DECREASED (Investigations) | 1 | 0
CACHEXIA (Metabolism and nutrition disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
ACUTE LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LIPOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MANTLE CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
MENINGIOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
HEMIANOPIA HETERONYMOUS (Nervous system disorders) | 1 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0
SEIZURE (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0
ANURIA (Renal and urinary disorders) | 0 | 1
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 | 0
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 1 | 0
OLIGURIA (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
OEDEMA GENITAL (Reproductive system and breast disorders) | 1 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 1 | 0
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 6 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
VOCAL CORD DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DRUG REACTION WITH EOSINOPHILIA AND SYSTEMIC SYMPTOMS (Skin and subcutaneous tissue disorders) | 1 | 0
HAEMORRHAGE (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 2 | 0
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=167) | Investigator's Choice (N=83)
ANAEMIA (Blood and lymphatic system disorders) | 45 | 18
LEUKOPENIA (Blood and lymphatic system disorders) | 29 | 18
LYMPHOPENIA (Blood and lymphatic system disorders) | 8 | 6
NEUTROPENIA (Blood and lymphatic system disorders) | 86 | 29
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 63 | 33
VERTIGO (Ear and labyrinth disorders) | 9 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 16 | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 | 6
CONSTIPATION (Gastrointestinal disorders) | 29 | 5
DIARRHOEA (Gastrointestinal disorders) | 36 | 8
DYSPEPSIA (Gastrointestinal disorders) | 9 | 3
NAUSEA (Gastrointestinal disorders) | 17 | 13
VOMITING (Gastrointestinal disorders) | 8 | 9
ASTHENIA (General disorders) | 26 | 11
FATIGUE (General disorders) | 34 | 4
OEDEMA PERIPHERAL (General disorders) | 16 | 9
PYREXIA (General disorders) | 26 | 9
BRONCHITIS (Infections and infestations) | 15 | 8
CONJUNCTIVITIS (Infections and infestations) | 9 | 0
INFLUENZA (Infections and infestations) | 9 | 1
NASOPHARYNGITIS (Infections and infestations) | 25 | 5
RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 23 | 5
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 22 | 3
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 9 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 15 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 16 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 13 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 13 | 0
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 0
HEADACHE (Nervous system disorders) | 14 | 0
PARAESTHESIA (Nervous system disorders) | 10 | 1
INSOMNIA (Psychiatric disorders) | 9 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 20 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10 | 6
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 9 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 15 | 3
RASH (Skin and subcutaneous tissue disorders) | 19 | 3
HYPERTENSION (Vascular disorders) | 15 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (4):
  • Study Protocol (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT00875667/Prot_000.pdf
  • Statistical Analysis Plan: CC-5013-MCL-002_SAP_Final_Redacted.19 December 2012 (2012-12-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT00875667/SAP_001.pdf
  • Statistical Analysis Plan: CC05013-MCL-002_SAP_2011_Redacted 18 July 2011 (2011-07-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT00875667/SAP_002.pdf
  • Statistical Analysis Plan: CC-5013-MCL-002_SAP_2010_Redacted 26 July 2010 (2010-07-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT00875667/SAP_003.pdf